CLINICAL TRIAL: NCT02979561
Title: A Prospective Randomised Controlled Study to Evaluate Outcomes of the Treatment With Pradaxa or Warfarin for Prevention of Recurrent VTE in Patients With Angiographically Confirmed Acute Massive Pulmonary Embolism Undergoing Endovascular Mechanical Fragmentation and Thrombolytic Therapy
Brief Title: Pradaxa or Warfarin for Prevention of Recurrent VTE in Patients With Angiographically Confirmed Acute Massive Pulmonary Embolism undergoIng Endovascular Mechanical Fragmentation and Thrombolytic Therapy
Acronym: Re-Spire
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RE-SPIRE study
Record Dates: First submitted 2016-11-22; First posted 2016-12-01 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-11

CONDITIONS: Angiographically Confirmed Acute Massive Pulmonary Embolism Treated With Endovascular Mechanical Fragmentation and Thrombolytic Therapy
Keywords: Dabigatran etexilate; Recurrence of DVT; Pulmonary Embolism; Warfarin
MeSH Terms: conditions — Pulmonary Embolism | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group of dabigatran (Experimental)
  Interventions: Drug: Dabigatran Etexilate
- group of warfarin (Active Comparator)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran Etexilate — All patients in this group continue to receive unfractionated heparin for 5-7 days, and then transferred to the drug Pradaxa dose of 150 mg 2 times a day. Pradaxa administration continued until the end of the treatment period. The treatment period starts on the day of randomization and lasts for 6 months.
  Arms: group of dabigatran
Drug: Warfarin — all patients continue to receive unfractionated heparin intravenously and at the same time (from the date of randomization) start warfarin, accompanied by regular measurement of the INR every day or every other day. As soon as INR reaches the range of 2.0 to 3.0, the administration of the unfractionated heparin should be discontinued. Further measurements of INR should be performed once a month during outpatient visits. The patient continues to receive warfarin under the control of the INR till the end of the treatment period. The treatment period starts on the day of randomization and lasts for 6 months.
  Arms: group of warfarin

SUMMARY:
A prospective randomised controlled study to evaluate outcomes of the treatment with pradaxa or warfarin for prevention of recurrent DVT in patients with angiographically confirmed acute massive pulmonary embolism undergoIng endovascular mechanical fragmentation and thrombolytic therapy. [RE-SPIRE study]

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged > 18 years
* Angiographically confirmed acute massive pulmonary embolism with involvement of Central pulmonary arteries.
* endovascular mechanical thrombus fragmentation + thrombolytic therapy (using recombinant tissue activator of plasminogen), performed for treatment of the above-mentioned pulmonary embolism in less than 48 hours before randomization. The patient should be randomized no earlier than 24 hours after procedures endovascular mechanical thrombus fragmentation + thrombolytic therapy
* Written informed consent signed by patient.

Exclusion Criteria:

* Signs of hemodynamic instability (i.e. systolic blood pressure <100 mm Hg.St. or episode of systolic blood pressure fall for ≥40 mm Hg. / or heart rate > 110 lasting more than 15 min) or need for ventilatory support within 12 hours prior to randomisation.
* The indication for oral anticoagulation, associated with others disease.
* malignant neoplasm of any location
* Contraindications to warfarin or pradaxa according to Russian Instructions for medical use of these drugs
* Indications for concomitant treatment with antiplatelet agents
* Any stroke within 6 months before randomization
* Intracranial hemorrhage in anamnesis
* Active bleeding, bleeding diathesis.
* Clinically significant bleeding within the last 30 days.
* Trauma or extensive surgery within 1 month before randomization or surgery planned in the next 6 months after randomization.
* Intracranial pathology: tumor, arteriovenous fistula or aneurysm.
* Gastrointestinal bleeding in the previous 3 months.
* Gastric ulcer or duodenal ulcer with clinical manifestations or endoscopically identified acute ulcer without signs of scarring during previous 30 days.
* Uncontrolled hypertension (systolic blood pressure> 180 mm Hg. and / or diastolic blood pressure> 100 mm.hg in patients receiving antihypertensive drugs).
* Pregnancy, lactation.
* Life expectancy <6 months.
* Clinically significant liver disease.
* Creatinine clearance (estimated by Cockcroft-Gault) <30 ml / min.
* hemoglobin level <90 g/l), thrombocytopenia <100x10^9 / L.
* Patients who, in the opinion of the researcher, are not suitable for inclusion in the study, for example, due to the low likelihood of doctor's recommendations following.
* Long-term use of NSAIDs
* Current participation in another clinical study.
* Allergic to contrast substance or radioisotope drugs used in procedures to assess endpoints of the study, which according to researchers, may be a contraindication to the implementation of these research methods.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
recurrent PE | 6 month
  according to Echocardiogram, scintigraphy of the lungs
death | 6 month

SECONDARY OUTCOMES:
hemorrhagic complications | 6 month
  according to the ISTH criteria
postembolic residual pulmonary hypertension | 6 month
  according to scintigraphy of the lungs
recurrent deep vein thrombosis | 3 month
  according to ultrasound of the deep veins
recurrent deep vein thrombosis | 6 month
  according to ultrasound of the deep veins

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Institution Academician E.N.Meshalkin Novosibirsk State Research Institute Of Circulation Pathology Rusmedtechnology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No